CLINICAL TRIAL: NCT02352506
Title: Macrophage Migration Inhibitory Factor in the Serum of Critically Ill Patients as an Early Marker for Acute Kidney Injury
Brief Title: Serum MIF in Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, David M Baron, MD, PhD, Univ.-Ass., Medical University of Vienna
Other Study IDs: 1680/2014
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum

GROUPS / COHORTS (2):
- AKI: Patients developing AKI during the ICU stay
  Interventions: Other: Blood draw for measurement of MIF
- No AKI: Matched controls not developing AKI during the ICU stay
  Interventions: Other: Blood draw for measurement of MIF

INTERVENTIONS:
Other: Blood draw for measurement of MIF — Observational study, no intervention

SUMMARY:
Acute kidney injury (AKI) is a common complication in critical care patients. Currently no parameters are available for early prognosis of AKI. Macrophage migration inhibitory factor (MIF) has been associated with AKI in clinical studies. The aim of this study is to evaluate the time course of MIF concentrations in patients with AKI.

ELIGIBILITY:
Exclusion Criteria:

* Age < 18 years and > 80 years
* Patients with chronic dialysis
* Patients with continuous hemodialysis, hemofiltration or hemodiafiltration within 4 weeks prior to the study
* Patients with an expected length of ICU stay shorter than 3 days
* Patients with a low probability of surviving the first 2 days after ICU admission
* Pregnancy and nursing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical care patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Macrophage migration inhibitory factor | Up to 14 days

SECONDARY OUTCOMES:
Serum creatinine | Up to 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria